CLINICAL TRIAL: NCT00520494
Title: A Multicenter Study on the Efficacy and Safety of Vivaglobin® in Previously Untreated Patients (PUPs) With Primary Immunodeficiency (PID)
Brief Title: Efficacy and Safety of Vivaglobin® in Previously Untreated Patients With Primary Immunodeficiency
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZLB06_005CR; 2006-006522-25 (EudraCT Number); 1461 (Other: CSL Behring)
Record Dates: First submitted 2007-08-23; First posted 2007-08-24 (Estimated); Results first posted 2013-05-03 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Common Variable Immunodeficiency; Agammaglobulinemia
Keywords: Previously Untreated Patient (PUP); Primary Immunodeficiency (PID); CVID; XLA; Subcutaneous immunoglobulin (SCIG); IgG trough level; Quality of life; Common variable immunodeficiency (CVID); X-linked agammaglobulinemia (XLA)
MeSH Terms: conditions — Common Variable Immunodeficiency; Agammaglobulinemia; Primary Immunodeficiency Diseases; Bruton type agammaglobulinemia | interventions — Vivaglobin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vivaglobin (Experimental): Vivaglobin: 16% (160 mg/mL) liquid formulation of human IgG for SC use. Loading dose: 100 mg/kg for 5 consecutive days; maintenance dose: 100 mg/kg 1 to 2 times a week for 24 weeks.
  Interventions: Drug: Vivaglobin

INTERVENTIONS:
Drug: Vivaglobin — Human normal immunoglobulin G (IgG) for subcutaneous (SC) use.

SUMMARY:
The objective of this study is to assess the efficacy and safety of Vivaglobin in previously untreated patients (PUPs) with primary immunodeficiency (PID) over a 25-week observation period. The purpose is to investigate whether PUPs will respond to subcutaneous immunoglobulin (SCIG) treatment with adequate trough levels without first receiving immunoglobulins by the intravenous route by demonstrating that 100 mg immunoglobulin G/kg body weight (IgG/kg bw) administered on 5 consecutive days (i.e. resulting in a total dose of 500 mg IgG/kg bw) results in an IgG increase to ≥ 5 g/L on Day 12 after initiation of SCIG therapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Written informed consent, age-adapted
* Male or female aged 1 to 70 years
* Diagnosis of primary humoral immunodeficiency
* No prior immunoglobulin substitution therapy
* IgG level of <5 g/L at screening
* Women of childbearing potential must use medically approved contraception and must have a negative urine pregnancy test at screening

Key Exclusion Criteria:

* Evidence of serious infection between screening and first treatment
* Bleeding disorders that require medical treatments
* Any medical disorder causing secondary immune disorders, autoimmune neutropenia, or a clinically significant defect in cell mediated immunity
* Any condition likely to interfere with evaluation of the study drug or satisfactory conduct of the trial

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Borte, MD, Principal Investigator — Klinik für Kinder-und Jugendmedizin am Städtischen Klinikum St. Georg, Leipzig, Germany
Locations (6):
- Canada (2):
  - Contact CSL Behring for facility details, Edmonton, Alberta
  - Contact CSL Behring for facility details, Montreal, Quebec
- Contact CSL Behring for facility details, Leipzig, Germany
- Italy (2):
  - Contact CSL Behring for facility details, Brescia
  - Contact CSL Behring for facility details, Roma
- Contact CSL Behring for facility details, Madrid, Spain

REFERENCES:
- [Result] Borte M, Quinti I, Soresina A, Fernandez-Cruz E, Ritchie B, Schmidt DS, McCusker C. Efficacy and safety of subcutaneous vivaglobin(R) replacement therapy in previously untreated patients with primary immunodeficiency: a prospective, multicenter study. J Clin Immunol. 2011 Dec;31(6):952-61. doi: 10.1007/s10875-011-9588-5. Epub 2011 Sep 20. PMID 21932110

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vivaglobin
Started | 18
Completed | 17
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vivaglobin
Number analyzed (Participants) | 18
Age Continuous [Mean (Standard Deviation); unit: years] | 25.9 (21.85)
Age, Customized [Number; unit: participants]
  2 to < 12 years | 6
  ≥ 12 to ≤ 16 years | 2
  > 16 to < 65 years | 8
  ≥ 65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10

OUTCOME MEASURES:

1. Secondary Outcome: Proportion of Patients Achieving IgG Levels ≥ 5 g/L on Day 19
Time Frame: On Day 19
Population: The ITT data set comprised all patients who were treated with the study drug and completed Day 12.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Vivaglobin
Number analyzed (Participants) | 18
proportion of participants | 0.944 [0.7271 to 0.9986]

2. Secondary Outcome: Proportion of Patients Achieving IgG Levels ≥ 5 g/L on Day 26
Time Frame: On Day 26
Population: The ITT data set comprised all patients who were treated with the study drug and completed Day 12.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Vivaglobin
Number analyzed (Participants) | 18
proportion of participants | 1.000 [0.8147 to 1.0000]

3. Secondary Outcome: IgG Increase (Change From Baseline) on Day 12
Time Frame: Baseline to Day 12
Population: The analysis population comprised all patients who were treated with the study drug and completed Day 12 (the ITT data set) and for which IgG results, as required for the analysis, were available.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Vivaglobin
Number analyzed (Participants) | 17
g/L | 3.941 (0.7466)

4. Secondary Outcome: Overall Rate of Infections
Description: Annualized rate of any infection. The annualized rate was based on the total number of infections and the total number of patient study days for all patients in the specified analysis population and adjusted to 365 days.
  Infections were classified as all AEs with the system organ class "infections and infestations".
Time Frame: For the duration of the study, up to approximately 25 weeks
Population: The ITT data set comprised all patients who were treated with the study drug and completed Day 12.
Measure: Number (95% Confidence Interval); unit: infections per patient year
Units Other Than Participants: Infections
Arm/Group | Vivaglobin
Number analyzed (Participants) | 18
Number analyzed (Infections) | 24
infections per patient year | 2.785 [1.785 to 4.144]

5. Secondary Outcome: Total Serum IgG Trough Levels on Day 12
Time Frame: On Day 12
Population: The ITT data set comprised all patients who were treated with the study drug and completed Day 12.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Vivaglobin
Number analyzed (Participants) | 18
g/L | 7.466 (1.4592)

6. Secondary Outcome: Total Serum IgG Trough Levels at Week 25
Time Frame: At Week 25
Population: The analysis population comprised all patients who were treated with the study drug and completed Day 12 (the ITT data set) and for which Week 25 total serum IgG results were available.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Vivaglobin
Number analyzed (Participants) | 17
g/L | 8.039 (1.1793)

7. Secondary Outcome: Serum Concentrations of Specific IgGs Against Cytomegalovirus, Tetanus, and Measles on Day 12
Time Frame: On Day 12
Population: The analysis population comprised all patients who were treated with the study drug and completed Day 12 (the ITT data set) and for which Day 12 specific IgG results were available.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Vivaglobin
Number analyzed (Participants) | 16
IU/mL
  Cytomegalovirus | 3.182 (0.8025)
  Tetanus | 1.399 (0.3846)
  Measles | 0.743 (0.3681)

8. Primary Outcome: Proportion of Patients Achieving Immunoglobulin G (IgG) Levels ≥ 5 g/L on Day 12
Time Frame: On Day 12
Population: The intention-to-treat (ITT) data set comprised all patients who were treated with the study drug and completed Day 12.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Vivaglobin
Number analyzed (Participants) | 18
proportion of patients | 0.944 [0.7271 to 0.9986]

9. Secondary Outcome: Serum Concentrations of Specific IgGs Against Cytomegalovirus, Tetanus, and Measles at Week 25
Time Frame: At Week 25
Population: The analysis population comprised all patients who were treated with the study drug and completed Day 12 (the ITT data set) and for which Week 25 specific IgG results were available.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Vivaglobin
Number analyzed (Participants) | 15
IU/mL
  Cytomegalovirus | 3.638 (2.2649)
  Tetanus | 1.623 (0.9344)
  Measles | 0.879 (0.8993)

10. Secondary Outcome: Serum Concentrations of Specific IgGs Against H. Influenzae Type B and S. Pneumoniae On Day 12
Time Frame: On Day 12
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Vivaglobin
Number analyzed (Participants) | 16
mg/L
  H. influenzae | 1.023 (0.3141)
  S. pneumoniae | 18.588 (9.4659)

11. Secondary Outcome: Serum Concentrations of Specific IgGs Against H. Influenzae Type B and S. Pneumoniae at Week 25
Time Frame: At Week 25
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Vivaglobin
Number analyzed (Participants) | 15
mg/L
  H. influenzae | 1.671 (0.7796)
  S. pneumoniae | 26.985 (22.2594)

12. Secondary Outcome: Use of Antibiotics for Infection Prophylaxis and Treatment
Description: Number of patients. Medications were classified as antibiotics according to the anatomic therapeutic chemical code.
Time Frame: For the duration of the study, up to approximately 25 weeks
Population: The ITT data set comprised all patients who were treated with the study drug and completed Day 12.
Measure: Number; unit: participants
Arm/Group | Vivaglobin
Number analyzed (Participants) | 18
participants
  Prophylaxis | 1
  Treatment | 8

13. Secondary Outcome: Quality of Life as Measured by the Adapted Short Form-36 Health Survey (SF-36; Age ≥ 14 Years)
Description: The SF-36 is a 36-item questionnaire that measures generic health concepts that are relevant across age, disease, and treatment groups. The questions are grouped into eight domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Scores range from 0 to 100, with higher scores indicating a better health state.
Time Frame: At study completion, approximately Week 25
Population: The analysis population comprised all patients who were treated with the study drug and completed Day 12 (the ITT data set), and for which responses to the SF-36 questionnaire were available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vivaglobin
Number analyzed (Participants) | 10
units on a scale
  Physical functioning | 75.50 (33.948)
  Role-physical | 70.63 (37.038)
  Bodily pain | 65.60 (37.262)
  General health | 56.40 (27.097)
  Vitality | 54.40 (28.575)
  Social functioning | 80.00 (30.162)
  Role-emotional | 79.17 (33.158)
  Mental health | 74.50 (23.268)

14. Secondary Outcome: Quality of Life as Measured by the Child Health Questionnaire Parent Form-50 (CHQ-PF50; Age ≤ 13 Years)
Description: The CHQ-PF50 is a 50-item questionnaire that measures generic health concepts and is suitable for patients younger than 14 years of age. The questions are grouped into 15 domains: global health, physical functioning, role/social limitations - emotional/behavioral, role/social limitations - physical, bodily pain, behavior, global behavior, mental health, self esteem, general health perceptions, change in health, parental impact - emotional, parental impact - time, family activities, and family cohesion. Scores range from 0 to 100, with higher scores indicating a better health state.
Time Frame: At study completion, approximately Week 25
Population: The analysis population comprised all patients who were treated with the study drug and completed Day 12 (the ITT data set), and for which responses to the CHQ-PF50 questionnaire were available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vivaglobin
Number analyzed (Participants) | 8
units on a scale
  Global health | 82.50 (15.353)
  Physical functioning | 97.91 (4.135)
  Role/social limitations - emotional/behavioral | 100.00 (0.000)
  Role/social limitations - physical | 95.84 (11.773)
  Bodily pain | 82.50 (24.349)
  Behavior | 74.06 (13.899)
  Global behavior | 75.63 (12.939)
  Mental health | 83.13 (13.871)
  Self esteem | 90.64 (6.948)
  General health perceptions | 61.66 (22.791)
  Change in health | 84.38 (18.601)
  Parental impact - emotional | 64.58 (39.530)
  Parental impact - time | 88.90 (15.698)
  Family activities | 86.98 (17.457)
  Family cohesion | 77.50 (15.353)

15. Secondary Outcome: Number of Patients With Adverse Events (AEs) by Severity and Relatedness
Description: Mild AE: Did not interfere with activities; Moderate AE: Interfered somewhat with routine activities; Severe AE: Impossible to perform routine activities.
  Not related: Explained by factors not involving the drug, no temporal relationship; Possibly related: Occurred within a reasonable time of administration, could also be explained by concurrent disease or other drugs; Probably related: Compelling temporal relationship, could not be explained concurrent disease/other drugs; Related AE: Compelling temporal relationship, known/suspected response to the drug confirmed by improvement on stopping.
Time Frame: For the duration of the study, up to approximately 25 weeks
Population: The Safety data set (SDS) comprised all treated patients.
Measure: Number; unit: participants
Arm/Group | Vivaglobin
Number analyzed (Participants) | 18
participants
  Total AEs | 14
  Mild AEs | 14
  Moderate AEs | 5
  Severe AEs | 2
  Not related AEs | 14
  Possibly related AEs | 3
  Probably related AEs | 4
  Related AEs | 5

16. Secondary Outcome: Rate of AEs by Severity and Relatedness
Description: The rate was the number of AEs over the number of infusions administered.
  Mild AE: Did not interfere with activities; Moderate AE: Interfered somewhat with routine activities; Severe AE: Impossible to perform routine activities.
  Not related: Explained by factors not involving the drug, no temporal relationship; Possibly related: Occurred within a reasonable time of administration, could also be explained by concurrent disease or other drugs; Probably related: Compelling temporal relationship, could not be explained concurrent disease/other drugs; Related AE: Compelling temporal relationship, known/suspected response to the drug confirmed by improvement on stopping.
Time Frame: For the duration of the study, up to approximately 25 weeks
Population: The SDS comprised all treated patients.
Measure: Number; unit: AEs per infusion
Units Other Than Participants: Infusions
Arm/Group | Vivaglobin
Number analyzed (Participants) | 18
Number analyzed (Infusions) | 551
AEs per infusion
  Total AEs | 0.305
  Mild AEs | 0.263
  Moderate AEs | 0.034
  Severe AEs | 0.007
  Not related AEs | 0.200
  Possibly related AEs | 0.013
  Probably related AEs | 0.018
  Related AEs | 0.074

17. Secondary Outcome: Number of Patients With Local Reactions by Severity and Relatedness
Description: Local reactions included: infusion site erythema, infusion site pain, infusion site pruritus, infusion site rash, infusion site reaction, infusion site swelling, injection site bruising, injection site erythema, injection site irritation, injection site pruritus, injection site swelling, edema peripheral, tenderness, erythema, pruritus, and skin swelling.
  Mild AE: Did not interfere with activities; Moderate AE: Interfered somewhat with routine activities; Severe AE: Impossible to perform routine activities.
  Not related: Explained by factors not involving the drug, no temporal relationship; Possibly related: Occurred within a reasonable time of administration, could also be explained by concurrent disease or other drugs; Probably related: Compelling temporal relationship, could not be explained concurrent disease/other drugs; Related AE: Compelling temporal relationship, known/suspected response to the drug confirmed by improvement on stopping.
Time Frame: For the duration of the study, up to approximately 25 weeks
Population: The SDS comprised all treated patients.
Measure: Number; unit: participants
Arm/Group | Vivaglobin
Number analyzed (Participants) | 18
participants
  Total local reactions | 6
  Mild local reactions | 6
  Moderate local reactions | 0
  Severe local reactions | 0
  Not related local reactions | 1
  Possibly related local reactions | 0
  Probably related local reactions | 1
  Related local reactions | 5

18. Secondary Outcome: Rate of Local Reactions by Severity and Relatedness
Description: The rate was the number of local reactions over the number of infusions administered.
  Local reactions included:
  * infusion site: erythema, pain, pruritus, rash, reaction, swelling;
  * injection site: bruising, erythema, irritation, pruritus, swelling;
  * edema peripheral;
  * tenderness;
  * erythema;
  * pruritus; and
  * skin swelling.
  Mild AE: Did not interfere with activities; Moderate AE: Interfered somewhat with routine activities; Severe AE: Impossible to perform routine activities.
  Not related: Explained by factors not involving the drug, no temporal relationship; Possibly related: Occurred within a reasonable time of administration, could also be explained by concurrent disease or other drugs; Probably related: Compelling temporal relationship, could not be explained concurrent disease/other drugs; Related AE: Compelling temporal relationship, known/suspected response to the drug confirmed by improvement on stopping.
Time Frame: For the duration of the study, up to approximately 25 weeks
Population: The SDS comprised all treated patients.
Measure: Number; unit: local reactions per infusion
Units Other Than Participants: infusions
Arm/Group | Vivaglobin
Number analyzed (Participants) | 18
Number analyzed (infusions) | 551
local reactions per infusion
  Total local reactions | 0.076
  Mild local reactions | 0.076
  Moderate local reactions | 0.000
  Severe local reactions | 0.000
  Not related local reactions | 0.004
  Possibly related local reactions | 0.000
  Probably related local reactions | 0.009
  Related local reactions | 0.064

19. Secondary Outcome: Number of Patients With Clinically Relevant Changes in Routine Laboratory Parameters
Description: Laboratory parameters included hematology, serum chemistry, and urinalysis parameters, and were assessed at screening, Week 12 (hematology and serum chemistry) and at the completion visit (approximately Week 25).
Time Frame: At Weeks 12 and 25
Population: The SDS comprised all treated patients.
Measure: Number; unit: participants
Arm/Group | Vivaglobin
Number analyzed (Participants) | 18
participants | 0

20. Secondary Outcome: Number of Patients With Clinically Relevant Changes in Vital Signs
Description: Vital signs included heart rate, systolic blood pressure, diastolic blood pressure, and body temperature.
Time Frame: At the screening visit, before and after infusions (Days 1 to 5), and at the completion visit (Week 25)
Population: The SDS comprised all treated patients.
Measure: Number; unit: participants
Arm/Group | Vivaglobin
Number analyzed (Participants) | 18
participants | 0

ADVERSE EVENTS:
Time Frame: For the duration of the study, up to approximately 25 weeks
Description: The SDS comprised all treated patients. Adverse events in "General disorders" were collected under the MedDRA System Organ Class (SOC) General disorders and administration site conditions.
Arm/Group | Vivaglobin
Serious Adverse Events (participants affected / at risk) | 2/18
Other Adverse Events (participants affected / at risk) | 14/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vivaglobin (N=18)
Headache (Nervous system disorders) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1)
Haemophilus infection (Infections and infestations) | 1 (1)
Pseudomonas bronchitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vivaglobin (N=18)
Nausea (Gastrointestinal disorders) | 4 (6)
Vomiting (Gastrointestinal disorders) | 2 (2)
Asthenia (General disorders) | 3 (3)
Fatigue (General disorders) | 2 (3)
Infusion site erythema (General disorders) | 2 (7)
Infusion site pain (General disorders) | 2 (4)
Injection site bruising (General disorders) | 2 (2)
Injection site erythema (General disorders) | 3 (5)
Injection site pruritus (General disorders) | 2 (3)
Injection site swelling (General disorders) | 4 (9)
Oedema peripheral (General disorders) | 2 (3)
Pyrexia (General disorders) | 5 (11)
Nasopharyngitis (Infections and infestations) | 2 (5)
Upper respiratory tract infection (Infections and infestations) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 5 (13)
Erythema (Skin and subcutaneous tissue disorders) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Haemolysis (Blood and lymphatic system disorders) | 1 (1)
Eye swelling (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (2)
Oral pain (Gastrointestinal disorders) | 1 (1)
Stomach discomfort (Gastrointestinal disorders) | 1 (1)
Swollen tongue (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Feeling hot (General disorders) | 1 (1)
Infusion site pruritus (General disorders) | 1 (1)
Infusion site rash (General disorders) | 1 (1)
Infusion site reaction (General disorders) | 1 (1)
Infusion site swelling (General disorders) | 1 (3)
Injection site irritation (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Tenderness (General disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (2)
Candidiasis (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (2)
Gastroenteritis (Infections and infestations) | 1 (3)
Otitis media (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (2)
Sinusitis (Infections and infestations) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (4)
Blood creatinine increased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2)
Disturbance in attention (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Nervousness (Psychiatric disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Renal pain (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus generalized (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1)
Skin swelling (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.